CLINICAL TRIAL: NCT05111847
Title: Safety and Performance of Short- and Long-term Baseplates for Attaching the UNEEG Episight Recorder- Part I
Brief Title: Safety and Performance of Short- and Long-term Baseplates for Attaching the UNEEG Episight Recorder - Part I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: U009 Part I
Record Dates: First submitted 2021-10-07; First posted 2021-11-08 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: In Part I of the study, the baseplates type A, B, C and D were tested on the skin behind the ears. Each subject tested either 1) short-term baseplates A and B first for 17/18 days and then long-term baseplates C and D for 17/18 days or 2) long-term baseplates C and D first for 17/18 days and then short-term baseplates A and B for 17/18 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term Baseplates first then long-term Baseplates (Other): Short-term Baseplates - Type A: Acrylate Type B: YUKI-gel
  Long-term Baseplates - Type C: Hydrocolloid Type D: Silicone
  Interventions: Device: Short-term Baseplates first then long-term Baseplates
- Long-term Baseplates first then short-term Baseplates (Other): Long-term Baseplates - Type C: Hydrocolloid Type D: Silicone
  Short-term Baseplates - Type A: Acrylate Type B: YUKI-gel
  Interventions: Device: Long-term Baseplates first then short-term Baseplates

INTERVENTIONS:
Device: Short-term Baseplates first then long-term Baseplates — Short-term Baseplates A and B tested for 17/18 days first then long-term Baseplates C and D tested for 17/18 days
  Arms: Short-term Baseplates first then long-term Baseplates
Device: Long-term Baseplates first then short-term Baseplates — Long-term Baseplates C and D tested for 17/18 days first then short-term Baseplates A and B tested for 17/18 days
  Arms: Long-term Baseplates first then short-term Baseplates

SUMMARY:
The purpose of this clinical investigation is to test the safety and performance of short- and longterm Baseplates constructed with different types of biocompatible adhesives.

DETAILED DESCRIPTION:
This clinical investigation intended to test different biocompatible adhesives over time as part of the UNEEG Episight Baseplate construction for UNEEG™ medical A/S

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained, and letter of authority signed before any study related activities
* Are at least 18 years of age and have full legal capacity
* Healthy skin behind the ear

Exclusion Criteria:

* Pregnant or breastfeeding
* Known allergic responses to the adhesives
* Treatment with corticosteroids, either as a cream in the area behind the ear or systemically (tablet or injection) within the last month
* Subject is unable or does not have the necessary assistance to properly operate the device system

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Karlsmark, Dr., Study Chair — Bispebjerg Hospital
Locations (1):
- Dermato-Venerologisk Afdeling og Videncenter for Sårheling, Bispebjerg Hospital, København NV, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was enrolled by mistake (and signed informed consent) but was immediately excluded.
  The subject was enrolled despite having a high degree of dandruff and thus did not have healthy skin as required per the inclusion criteria. This subject was not randomized and did not provide any data.
Units Other Than Participants: Head sides
Groups:
- Short-term Baseplates First, Then Long-term Baseplates: Started with 1-day use adhesives for 17-18 days:
  Type A: Acrylate behind one ear and Type B: YUKI-gel behind the other ear.
  Subsequently tested 4-days use adhesives for 17-18 days:
  Type C: Hydrocolloid behind one ear and Type D: Silicone behind the other ear
- Long-term Baseplates First, Then Short-term Baseplates: Started with 4-days use adhesives for 17-18 days:
  Type C: Hydrocolloid behind one ear and Type D: Silicone behind the other ear.
  Subsequently tested 1-day use adhesives for 17-18 days:
  Type A: Acrylate behind one ear and Type B: YUKI-gel behind the other ear.
Period: First intervention (17-18 days)
Arm/Group | Short-term Baseplates First, Then Long-term Baseplates | Long-term Baseplates First, Then Short-term Baseplates
Started | 16; 32 Head sides | 17; 34 Head sides
Completed | 15; 30 Head sides | 16; 32 Head sides
Not Completed | 1; 2 Head sides | 1; 2 Head sides
Period: Second intervention (17-18 days)
Arm/Group | Short-term Baseplates First, Then Long-term Baseplates | Long-term Baseplates First, Then Short-term Baseplates
Started | 15; 30 Head sides | 16; 32 Head sides
Completed | 14; 28 Head sides | 16; 32 Head sides
Not Completed | 1; 2 Head sides | 0; 0 Head sides

BASELINE CHARACTERISTICS:
Population: All enrolled participants in compliance with in- and exclusion criteria
Units Other Than Participants: Head sides
Groups:
- Total: Total of all reporting groups
Arm/Group | Short-term Baseplates First, Then Long-term Baseplates | Long-term Baseplates First, Then Short-term Baseplates | Total
Number analyzed (Participants) | 16 | 17 | 33
Number analyzed (Head sides) | 32 | 34 | 66
Age, Continuous [Median (Full Range); unit: years] — Population: All enrolled participants in compliance with in- and exclusion criteria
  years | 24.5 [20 to 71] | 45 [22 to 75] | 32 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All enrolled participants in compliance with in- and exclusion criteria
  Participants
    Female | 7 | 11 | 18
    Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All enrolled participants in compliance with in- and exclusion criteria
  Participants
    Hispanic or Latino | 2 | 0 | 2
    Not Hispanic or Latino | 12 | 17 | 29
    Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All enrolled participants in compliance with in- and exclusion criteria
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 10 | 16 | 26
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Trans Epidermal Water Loss (TEWL) to Measure Skin-friendliness
Description: To evaluate the skin barrier functionality (i.e., skin-friendliness) after repeated use of Baseplates (i.e., adhesives) on the skin behind the ear.
  High levels of TEWL reflects unhealthy skin, i.e. high loss of water that passes from inside a body through the epidermis.
Time Frame: 17-18 days
Population: Participants with at least one TEWL measurement following use of the given baseplate type
Measure: Mean (Standard Deviation); unit: g/m²/h
Units Other Than Participants: Head sides
Groups:
- Short-term Baseplate Type A: Acrylate: Short-term Baseplate type A tested behind one ear for 17-18 days
- Short-term Baseplate Type B: YUKI-gel: Short-term Baseplate type B tested behind one ear for 17-18 days
- Long-term Baseplate Type C: Hydrocolloid: Long-term Baseplate type C tested behind one ear for 17-18 days
- Long-term Baseplate Type D: Sillicone: Long-term Baseplate type D tested behind one ear for 17-18 days
Arm/Group | Short-term Baseplate Type A: Acrylate | Short-term Baseplate Type B: YUKI-gel | Long-term Baseplate Type C: Hydrocolloid | Long-term Baseplate Type D: Sillicone
Number analyzed (Participants) | 32 | 32 | 33 | 33
Number analyzed (Head sides) | 32 | 32 | 33 | 33
g/m²/h
  Test area | 20.7 (11.1) | 8.0 (2.4) | 19.3 (8.0) | 8.0 (3.0)
  Control area | 7.5 (2.1) | 7.3 (1.8) | 7.5 (1.8) | 7.1 (2.3)

2. Secondary Outcome: Skin Reactions
Description: Systematic assessment (visual inspection by investigator and self-reporting by participant via daily questionnaires). Some skin reactions were also reported as adverse device effects (see Adverse Event section)
Time Frame: 17-18 days
Population: Participants with at least one skin assessment after use of the given Baseplate type
Measure: Number; unit: Head sides
Units Other Than Participants: Head sides
Groups:
- Long-term Baseplate Type D: Silicone: Long-term Baseplate type D tested behind one ear for 17-18 days
Arm/Group | Short-term Baseplate Type A: Acrylate | Short-term Baseplate Type B: Yuki-gel | Long-term Baseplate Type C: Hydrocolloid | Long-term Baseplate Type D: Silicone
Number analyzed (Participants) | 32 | 32 | 33 | 33
Number analyzed (Head sides) | 32 | 32 | 33 | 33
Head sides | 24 | 15 | 29 | 26

ADVERSE EVENTS:
Time Frame: From enrollment until follow-up, 35-42 days. Each baseplate type tested for 17-18 days.
Description: Adverse device effects (ADEs) were categorized according to International Medical Device Regulators Forum (IMDRF). Skin reactions reported by visual inspection and daily questionnaires were also collected as a secondary endpoint separate from adverse event registration (see Outcome Measures).
Groups:
- Short-term Baseplate Type A: Acrylic: Short-term Baseplate type A tested behind one ear for 17-18 days
Arm/Group | Short-term Baseplate Type A: Acrylic | Short-term Baseplate Type B: Yuki-gel | Long-term Baseplate Type C: Hydrocolloid | Long-term Baseplate Type D: Silicone
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 22/32 | 15/32 | 29/33 | 26/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short-term Baseplate Type A: Acrylic (N=32) | Short-term Baseplate Type B: Yuki-gel (N=32) | Long-term Baseplate Type C: Hydrocolloid (N=33) | Long-term Baseplate Type D: Silicone (N=33)
Skin reaction (Skin and subcutaneous tissue disorders) | 22 | 14 | 29 | 26
Discomfort, pain, headache (General disorders) | 1 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
The study did not have a formal power and sample size calculation. Some skin reactions were reported both as an ADE and separately in the "skin reaction questionnaire".

When recording objective skin measurements, particularly TEWL, it is important that the room conditions, such as temperature and humidity, which may have affected the skin measurements. However, all TEWL measurements were within acceptable range.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT05111847/Prot_000.pdf